CLINICAL TRIAL: NCT03935763
Title: A Real World Evidence Prospective Cohort Study in the Management of Metastatic Colorectal Cancer: A Clinical and Patient Perspective
Brief Title: Management of Metastatic Colorectal Cancer: A Clinical and Patient Perspective
Acronym: PROMETCO
Status: Active, not recruiting | Type: Observational
Sponsor: Servier Affaires Médicales (Industry)
Responsible Party: Sponsor
Organization: Servier (Industry)
Other Study IDs: DIM-95005-001; EUPAS33865 (Other: EU PAS Register Number)
Record Dates: First submitted 2019-04-24; First posted 2019-05-02 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Real Worl Evidence
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: observational disease study — observation of routine clinical practices in mCRC

SUMMARY:
A Real World Evidence Prospective Cohort Study in the Management of Metastatic Colorectal Cancer: A Clinical and Patient Perspective

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Diagnosis of mCRC
* Having had two disease progressions since diagnosis of first metastasis that led to first systemic treatment.

Exclusion Criteria:

* Currently participating in an investigational clinical trial (thus it does not apply to observational cohort studies)
* Currently being treated for other cancer(s)
* Not having mental capacity and/or ability to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population will be adults with mCRC who are eligible and willing to receive subsequent treatment, having had two prior progressions since diagnosis of first metastasis.
Sampling Method: Non-Probability Sample
Enrollment: 738 (Actual)
Dates: Start 2019-03-08 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Overall survival | From date of randomization until the date of death from any cause, assessed up to 24 months months
  metastatic Colorectal Cancer (mCRC) overall survival in real world setting

SECONDARY OUTCOMES:
Disease control measured by overall response | within 18 months from enrollment
  Overall response to treatment defined by complete and partial response, stable disease, progression of the disease
Quality of life using Patients Reported Outcomes | within 18 months from enrollment
  Patients Reported Outcomes defined by a modified version of the questionnaire ACCEPTance by the Patients of their Treatment (ACCEPT)

CONTACTS AND LOCATIONS:
Locations (18):
- Instituto de Oncología Angel H. Roffo, Buenos Aires, Argentina
- Landeskrankenhaus-Universitaetsklinik, Salzburg, Austria
- Antwerp University Hospital, Edegem, Belgium
- Klinicki Bolnicki Centar (KBC) Zagreb, Zagreb, Croatia
- University Hospital in Hradec Kralove Clinic of Oncology and Radiotherapy, Hradec Králové, Czechia
- Groupe Hospitalier Pitié Salpêtrière, Paris, France
- Klinikum Wolfsburg, Wolfsburg, Germany
- University Hospital Of Heraklion, Heraklion, Greece
- Del-Pesti Centrum Korhaz OHII, Szent Laszlo Korhaz Telephely, Budapest, Hungary
- The Adelaide & Meath Hospital-Dublin Incorporating The National Children's Hospital, Dublin, Ireland
- Arcispedale Santa Maria Nuova, Reggio Emilia, Italy
- UMC Utrecht, Utrecht, Netherlands
- Centro Des Estudos Egas Moniz - Hospital Santa Maria, Lisbon, Portugal
- Institute Of Oncology Ljubljana, Ljubljana, Slovenia
- Hospital Universitario 12 de Octubre, Madrid, Spain
- Vasteras Central Hospital, Västerås, Sweden
- UniversitaetsSpital Zuerich (University Hospital Zurich), Zurich, Switzerland
- Cancer Research UK, Department of Medical Oncology-The Christie NHS Foundation Trust, Manchester, United Kingdom

REFERENCES:
- [Derived] Moss B, Goodall EA, Maravic Z, Marti F, Moss M, Rowley S, Sarrauste C, Wheatstone P. Real-world evidence research in metastatic colorectal cancer: raising awareness of the need for patient contributions. Future Oncol. 2023 Aug;19(26):1809-1821. doi: 10.2217/fon-2022-1253. Epub 2023 Jul 13. PMID 37439564
- [Derived] Koopman M, Pinto C, Bodoky G, Garcia-Carbonero R, Marti FM, Bachet JB. Rationale and design of the PROMETCO study: a real-world, prospective, longitudinal cohort on the continuum of care of metastatic colorectal cancer from a clinical and patient perspective. Future Oncol. 2022 Apr;18(11):1313-1320. doi: 10.2217/fon-2021-1333. Epub 2022 Jan 19. PMID 35043682